CLINICAL TRIAL: NCT06370572
Title: Pragmatic Use of PAIN-Advanced Dementia Scale in Emergency Departments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIRB23-1162; U54AG063546 (NIH)
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-06

CONDITIONS: Dementia; Hip Pain; Emergency Department Patient; Pain in Advanced Dementia Scale
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This is a interrupted time series intervention, which allows a pre- and post-intervention assessment of the effect of PAINAD scale.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-implementation (No Intervention): PLWD presenting to the ED with reported hip pain in the year preceding implementation of the PAINAD EHR prompt
- Post-implementation (Experimental): PLWD presenting to the ED with reported hip pain in the 10 months following implementation of the PAINAD EHR prompt
  Interventions: Other: PAINAD EHR Prompt

INTERVENTIONS:
Other: PAINAD EHR Prompt — Implementation of PAINAD EHR prompt in the ED workflow for PLWD presenting to the ED with hip pain
  Arms: Post-implementation

SUMMARY:
The purpose of this study is to learn if the Pain in Advanced Dementia (PAINAD) scale can improve emergency pain care in persons living with dementia (PLWD). It is hypothesized that a PAINAD electronic health record (EHR) prompt that appears to emergency department (ED) staff will enable them to accurately assess pain levels and lead to better pain treatment for PLWD.

DETAILED DESCRIPTION:
This is a pragmatic pilot for a Stage IV effectiveness, embedded pragmatic clinical trial (ePCT) studying the feasibility of PAINAD assessment implementation via simple EHR prompts for PLWD presenting to the ED with hip pain at the University of Chicago Medicine (UCM) and the University of North Carolina at Chapel Hill (UNC-CH). Identification of subjects with hip pain and dementia contains the level of specificity needed for a pragmatic trial, and occurs on ED arrival, prompting an electronic health record clinical decision support (CDS).

The Pain in Advance Dementia (PAINAD) Score is a behavioral score based on observation of the person. The score depends on observation of five behaviors, breathing, negative vocalizations, facial expressions, body language, and consolability. Each observed behavior is scored from zero = none, to two = most, for a total score from zero to ten.

The design is an interrupted time series intervention, which allows a pre- and post-intervention assessment of the effect of PAINAD scale. Pre-intervention data from most immediate year to date prior to the intervention start defines the baseline state. The intervention, the EHR prompt to document the PAINAD first on patient arrival to the ED treatment area, and second one hour after delivery of first pain treatment. Prospective evaluation of EHR data will be used to evaluate use of the PAINAD.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 65 years old
* ED arrival complaint of hip pain
* History of dementia by past medical history or problem list in EHR

Exclusion Criteria:

* Patients do not meet inclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 714 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible patients receiving a PAINAD assessment upon ED arrival | 10 months post-implementation of PAINAD CDS in the ED
  Measured by numbers of patients

SECONDARY OUTCOMES:
Change in time to administration of first analgesic medication | Baseline (end of 1 year preceding implementation), 10 months
  Measured by length of time in minutes
Change in pain score for patients receiving a repeat PAINAD assessment | Baseline (end of 1 year preceding implementation), 10 months
  Measured by PAINAD score; scores range from 0 to 10 (based on a scale of 0 to 2 for five items), with a higher score indicating more severe pain (0="no pain" to 10="severe pain")

CONTACTS AND LOCATIONS:
Overall Officials: Teresita M Hogan, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina